CLINICAL TRIAL: NCT06718244
Title: A Clinical Study of Inaticabtagene Autoleucel (Inati-cel; CNCT19) Treatment for B-Cell Acute Lymphoblastic Leukemia(B-ALL) Patients in First Complete Remission (CR1)，Minimal Residual Disease(MRD) Positive
Brief Title: Inaticabtagene Autoleucel (Inati-cel; CNCT19) Treatment for MRD-Positive B-ALL Patients in CR1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jin Wang, chief physician, MD, PhD, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (2024) Ruijin Ethics No.447
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Minimal Residual Disease; Chimeric Antigen Receptor T (CAR-T)Cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention group (Experimental): Administration with Inaticabtagene autoleucel CD19 CAR-T cells in the MRD positive B-ALL patients in CR1.
  Interventions: Biological: single dose of Inaticabtagene autoleucel

INTERVENTIONS:
Biological: single dose of Inaticabtagene autoleucel — Inaticabtagene autoleucel will be transfusioned intravenously at the recommended dose of 0.5×10^8 (ranging 0.2-0.6×10^8) viable CAR-T cells.
  If the quantity of CAR-T cells of the patient is sufficient, after the patient receives the first CAR-T transfusion 5~6 months，they will receive a second CAR-T cell transfusion. The aim of the second transfusion is to prolong the duration of CAR-T in the patient's body and prolong the patient's DOR. The dose and procedures of the second transfusion are the same as those for the first transfusion. After the second infusion, the patient will receive evaluation based on the day of the second transfusion as Day0.
  Other Names: Inati-cel; CNCT-19

SUMMARY:
This investigator-initiated, prospective, single-arm, open-label, single-center clinical study aims to evaluate the efficacy and safety of Inaticabtagene autoleucel (Inati-cel;CNCT19)CD19 CAR-T theraphy in adults B-ALL that are in first complete remission(CR1) with minimal residual disease (MRD) positivity. This trial will enroll 20 participants for leukapheresis and treatment with lymphodepleting chemotherapy followed by Inati-cel CAR T cell infusion. Patients will be assessed for MRD negativity rate(at months 1, 2, 3, and 6 after CAR-T transfusion), duration of MRD negativity, overall survival(OS), relapse-free survival(RFS), pharmacokinetics(PK) characteristics, incidence of adverse events(AEs), exploratory biomarker research at 1,2,3,6,9,12,15,18,21 and 24- months post Inati-cel infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥16 and ≤70 years at screening, no gender restrictions
* ECOG score of 0-1 at screening
* Newly diagnosed Ph-negative B-ALL, MRD positive(bone marrow MRD ≥0.01% by flow cytometry) in CR1 (with <5% blasts in bone marrow, no blasts in peripheral blood, no extramedullary disease)after induction chemotherapy or consolidation chemotherapy.
* Newly diagnosed Ph-positive B-ALL, MRD positive(bone marrow MRD ≥0.01% by flow cytometry or BCR-ABL1 >0.01% detected by qPCR) in CR1 (with <5% blasts in bone marrow, no blasts in peripheral blood, no extramedullary disease) .
* At diagnosis of B-ALL,CD19 expression of leukemic cells is positive by flow cytometry in bone marrow or peripheral blood.
* Appropirate organ function, meeting the following criteria:

  1. Aspartate aminotransferase (AST) ≤3 times the upper limit of normal (ULN);
  2. Alanine aminotransferase (ALT) ≤3 times ULN;
  3. Total bilirubin ≤2 times ULN (for patients with Gilbert's syndrome, total bilirubin ≤3.0 times ULN and direct bilirubin ≤1.5 times ULN);
  4. Serum creatinine ≤1.5 times ULN, or creatinine clearance ≥60 mL/min (using the Cockcroft-Gault formula);
  5. International Normalized Ratio (INR) ≤1.5 times ULN and activated partial thromboplastin time (APTT) ≤1.5 times ULN;
  6. Left ventricular ejection fraction (LVEF) ≥50%;
  7. Minimum pulmonary reserve, with oxygen saturation >91% on room air;
* Meets leukapheresis standard of the study center, with no contraindications for blood cell separation;
* Voluntarily agrees to participate in this study and signs on the informed consent form(ICF).

Exclusion Criteria:

* Received CAR-T cell therapy before screening;
* Inherited bone marrow failure syndrome(IBMFS) or any other known bone marrow failure syndromes;
* Active systemic autoimmune diseases requiring treatment;
* Any of the following conditions:

  1. HBsAg and/or HBeAg positive;
  2. HBe-Ab and/or HBc-Ab positive with HBV-DNA levels above the lower limit of quantification;
  3. HCV-Ab positive;
  4. TP-Ab positive;
  5. HIV antibody positive;
  6. EBV-DNA or CMV-DNA levels above the lower limit of quantification;
* Active infection at screening.
* Any other malignancy within the past five years before screening, excluding cases where the patient has been disease-free for more than 5 years after curative treatment or has a low risk of relapse as assessed by the investigator;
* Any of the following cardiac conditions:

  1. NYHA Class III or IV congestive heart failure;
  2. Severe arrhythmia requiring treatment;
  3. Uncontrolled hypertension or pulmonary hypertension despite standard therapy;
  4. Unstable angina;
  5. Myocardial infarction, bypass surgery, or stent placement within six months before cell retransfusion;
  6. Clinically significant valvular disease;
  7. Other cardiac conditions deemed unsuitable by the investigator;
* History of epilepsy, cerebellar disease, or other active central nervous system disorders;
* Uncontrolled diabetes;
* History of symptomatic deep vein thrombosis or pulmonary embolism within six months before screening that is not well controlled;
* History of hypersensitivity to any component of the investigational product.
* Received a live vaccine within six weeks before screening;
* Life expectancy of less than three months;
* Participation in another interventional clinical trial and receiving investigational drugs within three months (for unapproved drugs) or within five half-lives (for approved drugs) before cell infusion, or plans to participate in another clinical trial or receive anti-cancer therapy outside the study protocol during the study period;
* Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
MRD negativity rate | up to 24 months
  The proportion of patients who reach MRD negative.Bone marrow of every patient will be analysed by multiparameter flow cytometry or/and RT-qPCR for MRD evaluation.

SECONDARY OUTCOMES:
Duration of MRD negativity | till the end of the study, up to 5 years
  Time from the first assessment of MRD negative to the first assessment of MRD positive or death from any cause.Bone marrow of every patient will be analysed by multiparameter flow cytometry or/and RT-qPCR for MRD evaluation.
Relapse-free survival (RFS) | till the end of the study, up to 5 years
  Interval from the date of transfusion of the Inati-cel to the time of hematological recurrence or death from any cause. Evaluation of RFS will be based on follow-up results.
Overall survival (OS) | till the end of the study, up to 5 years
  Interval from the date of the feedback to the time of death due to any reason. Evaluation of OS will be based on follow-up results.
incidence of adverse events | up to 24 months
  The proportion of patients who have adverse events after Inati-cel transfusion.Adverse events will be assessed by CTCAE v5.0
Pharmacokinetics characteristics of Inati-cel | till the end of the study, up to 5 years
  Including duration of CAR T cells, relative proportion of CAR-T cells and absolute counts of CAR-T cells.These will be evaluated by multiparameter flow cytometry.
exploratory biomarker research | till the end of the study, up to 5 years
  A small amount of blood or bone marrow will be collected for further biomarker research, including flowcytometric analysis of lymphocyte subsets, multiomics analysis of leukenic cells and CAR-T cells, in vivo and in vitro experiments on drug interference in CAR-T therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No